CLINICAL TRIAL: NCT01902589
Title: Resistance of Helicobacter Pylori to Antibiotics in Children
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0058-10-EMC
Record Dates: First submitted 2011-09-27; First posted 2013-07-18 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Abdominal Pain; Children; Bacterial Infection Due to Helicobacter Pylori (H. Pylori); Antibiotic Resistant Strain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Helicobacter pilorii in biopsy: Patients with Helicobacter pylori in biopsy, cultures will be obtained and subsequently sensitivity to antibiotics studied.
  Interventions: Other: Helicobacter Pylori Culture

INTERVENTIONS:
Other: Helicobacter Pylori Culture — Biopsy specimens for histology will be fixed in formalin, embedded in paraffin and sectioned and stained with hematoxylin and eosin.
  The microbiological workup will include an imprint of the biopsy on a slide followed by a gram stain for the purpose of demonstrating H. pylori in situ. Further the biopsies will be streaked out on chocolate agar, Sheep blood agar and H. pylori selective agar supplemented with Polymixin to suppress possible contaminants.
  4 days of incubation in a micro aerophilic atmosphere will follow . Susceptibility testing of H pylori will be performed with E test on Mueller Hinton agar supplemented with defibrinated sheep blood using a MacFalrland 3.0 density of a bacterial suspension. Reading the susceptibility will take place following 72 hours of incubation in a micro aerophilic atmosphere.

SUMMARY:
Helicobacter Pylori (HP) is one of the most common pathogens in humans. This infection can present in children with abdominal pain, vomiting and iron deficiency. The treatment is usually empiric and includes antibiotic treatment usually Amoxycillin and Clarithromycin or Metronidazole. Between 40 to 70 % of the pathogens are resistant to those drugs, and it is important to characterize the specific sensitivity of the pathogens in any specific area and in pediatric population. The aims of this study is to assess the sensitivity of HP in pediatric population in Northern Israel.

DETAILED DESCRIPTION:
The aim of our prospective study is to investigate the rate of H pylori resistant strains to antibiotic treatment including Amoxicillin, Clarithromycin, Metronidazole, Tetracycline and Quinolones in pediatric population in Ha-Emek medical center, Afula. The second aim was to determine if in vitro resistance is being reflected in vivo too.

Should the investigators find high rates of H pylori resistance to Clarithromycin, the investigators will have to reconsider the recommendation to use Clarithromycin as the first line treatment for H pylori.

Our research group will conclude 100 children in the ages of 1-18 years, evaluated for recurrent abdominal pain, iron deficiency anemia, failure to thrive by an upper endoscopy, biopsy specimens taken for a rapid urease test, for histology, for culture and for antibiotic susceptibility testing.

Biopsy specimens for histology will be fixed in formalin, embedded in paraffin and sectioned and stained with hematoxylin and eosin.

The microbiological workup will include an imprint of the biopsy on a slide followed by a gram stain for the purpose of demonstrating H. pylori in situ. Further the biopsies will be streaked out on chocolate agar, Sheep blood agar and H. pylori selective agar supplemented with Polymixin to suppress possible contaminants.

4 days of incubation in a micro aerophilic atmosphere will follow . Susceptibility testing of H pylori will be performed with E test on Mueller Hinton agar supplemented with defibrinated sheep blood using a MacFalrland 3.0 density of a bacterial suspension. Reading the susceptibility will take place following 72 hours of incubation in a micro aerophilic atmosphere.

ELIGIBILITY:
Inclusion Criteria:

* ages of 1-18 years,
* evaluated for recurrent abdominal pain,
* iron deficiency anemia,
* failure to thrive by an upper endoscopy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our research group will conclude 100 children in the ages of 1-18 years, evaluated for recurrent abdominal pain, iron deficiency anemia, failure to thrive by an upper endoscopy, biopsy specimens taken for a rapid urease test, for histology, for culture and for antibiotic susceptibility testing.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Resistance of specific organism to antibiotics | Two weeks from the culture

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Peleg, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Ha'Emek Medical Center, Afula, Israel